CLINICAL TRIAL: NCT04897152
Title: Coronavirus Associated Pneumomediastinum and Pneumothorax - COVIMIX Study
Brief Title: Coronavirus Associated Pneumomediastinum and Pneumothorax
Acronym: COVI-MIX
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Clinical Professor in Anesthesiology and Intensive Care, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: COVI-MIX
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Pneumothorax; Pneumomediastinum; COVID-19 Pneumonia
MeSH Terms: conditions — Pneumothorax; Mediastinal Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spontaneous pneumomediastinum (PMS) is defined as free air within the mediastinum. Spontaneous pneumothorax (PNX) consists of the presence of air inside the pleural space. PMS and PNX may sometimes occur secondly to an underlying pathology, or deriving from a sudden increase in intra-alveolar pressure such as functional alteration such as airway hyperactivity, Valsalva maneuver, cough, barotrauma, and/or volutrauma with consequent rupture of the alveoli and subsequent leakage of air into the mediastinum due to the Macklin effect. The escaping air can then spread inside the pericardium, the peritoneum, the muscles, and subcutaneous tissues, hence causing subcutaneous emphysema.

PMS and PNX are rare complications of several lung infections such as Pneumocystis Jirovecii pneumonia, tuberculosis, bacterial necrotizing pneumonia, and herpes pneumonia.

However, an increasing number of PMS and PNX has been described in patients with SARS-CoV2 interstitial pneumonia. PMS and PNX can either present as the onset manifestation of COVID-19 disease, or occur as complications of non-invasive and/or invasive ventilation, or following to cystic and/or fibrotic evolution of the pathology.

The frequency of PMS and PNX during COVID-19 is not well defined, as the available data are limited to case collections and single reports. According to currently available scientific literature, PNX in COVID-19 occurs with frequency rates of 1-3%, up to 6% in patients undergoing non-invasive ventilation (NIV) and mechanical artificial ventilation (VAM). In McGuinness's analysis, which compared the complications of barotrauma in patients with acute respiratory distress syndrome (ARDS) in VAM, PNX and PMS occurred with frequency rates of 9% and 10%, respectively, while in non-COVID-19 population, PNX and PMS frequency rates were 12% and 3%, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older hospitalized with SARS-COV2 infection

Exclusion Criteria:

* Failure to obtain clinical or radiological information about the case

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with SARS-COV2 infection
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Barotrauma occurrence with different respiratory strategies | February 20, 2020 - March 31, 2021
  Effect of the different respiratory support strategies on barotrauma (pneumomediastinum and/or pneumothorax) occurrence

SECONDARY OUTCOMES:
Pneumomediastinum and pneumothorax | February 20, 2020 - March 31, 2021
  Estimating pneumomediastinum and pneumothorax frequency rates in hospitalized COVID-19 patients
Risk factors other than ventilation strategy | February 20, 2020 - March 31, 2021
  Evaluating risk factors associated with barotrauma (spontaneous breathing, non-invasive, invasive, or extracorporeal circulation) in hospitalized COVID-19 patients
30-day outcome | 30 days
  Assessment of the in-hospital outcome, intended as "survival days" in hospitalized COVID-19 patients who manifest barotrauma

CONTACTS AND LOCATIONS:
Locations (27):
- Italy (27):
  - Policlinico S.Orsola-Malpighi, Pneumologia e Terapia Intensiva Respiratoria, Bologna
  - Policlinico S.Orsola-Malpighi, U.O Malattie Infettive, Bologna
  - Azienda Ospedaliero-Universitaria V.Emanuele Ferrarotto, S.bambino, Malattie Infettive, Catania
  - Azienda Ospedaliero-Universitaria V.Emanuele Ferrarotto, S.bambino, U.O.C. di Malattie Infettive, Catania
  - Azienda Ospedaliera S.Croce e Carle Cuneo, SC Malattie Infettive e tropicali,, Cuneo
  - Ospedale Policlinico San Martino-IRCCS, Clinica di Malattie Infettive e Tropicali, Genova
  - Fondazione IRCCS, Ca Granda Ospedale Maggiore Policlinico, UOC, Malattie Infettive, Milan
  - Ospedale dei colli, Malattie Infettive ed Urgenze Infettivologiche,, Napoli
  - Azienda Ospedaliera di Padova, S.C di Fisiopatologia respiratoria,, Padua
  - Unità Operativa Complessa Istituto di Anestesia e Rianimazione dell'Azienda Ospedale-Università di Padova,, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone di Palermo, UOC Anestesia Rianimazione con Terapia Intensiva Polivalente e del Dolore, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Clinica Pneumologica, Parma
  - Azienda Ospedaliera Perugia, Malattie Infettive, Perugia
  - Azienda USL Toscana Ovest, Ospedale Felice Lotti SOC Medicina Interna, Pontedera
  - Azienda Sanitaria Universitaria Friuli Occidentale, S.C Pneumologia, Pordenone
  - AOU Città della Salute e Scienza, SC Malattie Infettive, Torino
  - Azienda Ospedaliera Ordine Mauriziano S.C. Pneumologia e Unità di Terapia Semi Intensiva Respiratoria, Torino
  - Ospedale Cardinal Massaia, SC Malattie Infettive, Torino
  - Azienda Sanitaria Universitaria Giuliano Isontina, S.C Pneumologia, Trieste
  - Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD, Udine
  - Azienda ospedaliero universitaria Friuli Centrale, Anestesia e Rianimazione 1, Udine
  - Azienda ospedaliero universitaria Friuli Centrale, Anestesia e Rianimazione 2, Udine
  - Azienda ospedaliero universitaria Friuli Centrale, Clinica di Anestesia e Rianimazione, Udine
  - Azienda Ospedaliero Universitaria Friuli Centrale, Malattie infettive, Udine
  - Azienda Ospedaliero Universitaria Friuli Centrale, Pneumologia, Udine
  - Azienda Sanitaria locale di Vercelli, Malattie infettive, Vercelli
  - Università di Verona, Clinica delle Malattie Infettive e Tropicali, Verona

REFERENCES:
- [Background] Maunder RJ, Pierson DJ, Hudson LD. Subcutaneous and mediastinal emphysema. Pathophysiology, diagnosis, and management. Arch Intern Med. 1984 Jul;144(7):1447-53. PMID 6375617
- [Background] Wang W, Gao R, Zheng Y, Jiang L. COVID-19 with spontaneous pneumothorax, pneumomediastinum and subcutaneous emphysema. J Travel Med. 2020 Aug 20;27(5):taaa062. doi: 10.1093/jtm/taaa062. PMID 32330274
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Yao W, Wang T, Jiang B, Gao F, Wang L, Zheng H, Xiao W, Yao S, Mei W, Chen X, Luo A, Sun L, Cook T, Behringer E, Huitink JM, Wong DT, Lane-Fall M, McNarry AF, McGuire B, Higgs A, Shah A, Patel A, Zuo M, Ma W, Xue Z, Zhang LM, Li W, Wang Y, Hagberg C, O'Sullivan EP, Fleisher LA, Wei H; collaborators. Emergency tracheal intubation in 202 patients with COVID-19 in Wuhan, China: lessons learnt and international expert recommendations. Br J Anaesth. 2020 Jul;125(1):e28-e37. doi: 10.1016/j.bja.2020.03.026. Epub 2020 Apr 10. PMID 32312571
- [Background] McGuinness G, Zhan C, Rosenberg N, Azour L, Wickstrom M, Mason DM, Thomas KM, Moore WH. Increased Incidence of Barotrauma in Patients with COVID-19 on Invasive Mechanical Ventilation. Radiology. 2020 Nov;297(2):E252-E262. doi: 10.1148/radiol.2020202352. Epub 2020 Jul 2. PMID 32614258
- [Derived] Vetrugno L, Castaldo N, Fantin A, Deana C, Cortegiani A, Longhini F, Forfori F, Cammarota G, Grieco DL, Isola M, Navalesi P, Maggiore SM, Bassetti M, Chetta A, Confalonieri M, De Martino M, Ferrari G, Francisi D, Luzzati R, Meini S, Scozzafava M, Sozio E, Tascini C, Bassi F, Patruno V; Italian COVI-MIX Study Group; De Robertis E, Aldieri C, Ball L, Baratella E, Bartoletti M, Boscolo A, Burgazzi B, Catalanotti V, Confalonieri P, Corcione S, De Rosa FG, De Simoni A, Bono VD, Tria RD, Forlani S, Giacobbe DR, Granozzi B, Labate L, Lococo S, Lupia T, Matellon C, Mehrabi S, Morosi S, Mongodi S, Mura M, Nava S, Pol R, Pettenuzzo T, Quyen NH, Rescigno C, Righi E, Ruaro B, Salton F, Scabini S, Scarda A, Sibani M, Tacconelli E, Tartaglione G, Tazza B, Vania E, Viale P, Vianello A, Visentin A, Zuccon U, Meroi F, Buonsenso D. Ventilatory associated barotrauma in COVID-19 patients: A multicenter observational case control study (COVI-MIX-study). Pulmonology. 2023 Nov-Dec;29(6):457-468. doi: 10.1016/j.pulmoe.2022.11.002. Epub 2022 Nov 24. PMID 36669936